CLINICAL TRIAL: NCT02765373
Title: Effects of Adjuvant Endocrine Therapy With Aromatase Inhibitors on the Postoperative Lipid Levels in Postmenopausal Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Principal Investigator, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CH-BC-030
Record Dates: First submitted 2016-04-08; First posted 2016-05-06 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: aromatase inhibitors; lipid levels
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Letrozole; Anastrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- steroidal aromatase inhibitors(AIs): Exemestane 25mg Qd for 5 years
  Interventions: Drug: Exemestane
- non-steroidal aromatase inhibitors(AIs): Letrozole 2.5mg Qd or Anastrozole 1mg Qd for 5 years
  Interventions: Drug: Letrozole; Drug: Anastrozole

INTERVENTIONS:
Drug: Exemestane
  Groups: steroidal aromatase inhibitors(AIs)
Drug: Letrozole
  Groups: non-steroidal aromatase inhibitors(AIs)
Drug: Anastrozole
  Groups: non-steroidal aromatase inhibitors(AIs)

SUMMARY:
This study is a prospective, controlled phase IV clinical trial among postmenopausal patients with hormone receptor-positive breast cancer.The main purpose is to compare the effects of steroidal aromatase inhibitor (AI) exemestane and non-steroidal AIs on the lipid levels of breast cancer patients.

DETAILED DESCRIPTION:
The study subjects are composed of postmenopausal women with hormone receptor-positive breast cancer who have received exemestane, anastrozole or letrozole followed by testing of safety variables such as low-density lipoprotein- cholesterol (LDL-C), triglyceride(TC), total cholesterol, high-density lipoprotein cholesterol(HDL), blood calcium, transaminase and fasting plasma glucose at different time intervals in two years.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic analysis verifies to be early-stage invasive breast cancer while immunohistochemistry shows estrogen receptor(ER) and/or progesterone receptor(PR) positive (ER/PR positive is defined that >1% of cells are positive).
2. The patients have received surgery for breast cancer and recovered well for an interval of at least 1 week.
3. The patients have received post-operational adjuvant chemotherapy and/or adjuvant radiotherapy whereas the interval of chemotherapy and/or adjuvant radiotherapy is more than 2 weeks.
4. The postmenopausal women have been confirmed to be to menopausal as defined in NCCN guidelines(including post bilateral oophorectomy; age≥60 year-old; age≤60 year-old, menopause for more than 1 year and plasma Follicle-Stimulating Hormone (FSH) and estradiol levels meet the menopausal scope).
5. Do not receive concomitant endocrine therapy, e.g. drug-induced menopause, tamoxifen.
6. The patients do not have severe cardiopulmonary dysfunction.
7. ECOG score: 0-1
8. The patients have enough organ function and meet the scope of aromatase inhibitors(AIs) therapy. The laboratory test indexes must comply with the following requirements:

   Blood routine: neutrophil≥1.5G/L, platelet count ≥75G/L, hemoglobin ≥100g/L Liver function: serum bilirubin ≤ 2 times the upper limit of normal value; ALT and AST≤3 times the upper limit of normal value; Renal function: serumcreatinine≤140μmol/L
9. Serum low density lipoprotein-cholesterol(LDL-C) value <3.37mmol/L
10. Imaging examination identifies none of local recurrence or distal metastasis.
11. No other combined malignancy.
12. The patients have good compliance to the therapy and follow-up to be scheduled and are able to understand the study protocol and sign the Informed Consent Form.

Exclusion criteria

1. The patients are not qualified to receive the adjuvant endocrine therapy with AIs.
2. The patients previously received other endocrine therapy (e.g. tamoxifen) simultaneity or the treatment with AIs (excluding those with a course of less than 3 months)
3. The patients received or are receiving the lipid-lowering therapy.
4. The patients suffer from other combined malignancy.
5. The patients have uncontrollable mental illness.
6. The patients experience severe cardiovascular diseases in the recent 6 months (e.g. unstable angina, chronic heart failure, uncontrollable hypertension >150/90 mmHg, myocardial infarction or cerebrovascular disorders).

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: postmenopausal women with hormone receptor-positive breast cancer who have received surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Ratio of patients whose low density lipoprotein-cholesterol（LDL-C） level ≥ 4.14 mmol/L in 2 years of administration among groups | Change of LDL-C level from Baseline to up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang X, Zhu A, Wang J, Ma F, Liu J, Fan Y, Luo Y, Zhang P, Li Q, Xu B, Yuan P. Steroidal aromatase inhibitors have a more favorable effect on lipid profiles than nonsteroidal aromatase inhibitors in postmenopausal women with early breast cancer: a prospective cohort study. Ther Adv Med Oncol. 2020 May 26;12:1758835920925991. doi: 10.1177/1758835920925991. eCollection 2020. PMID 32518597